CLINICAL TRIAL: NCT06253156
Title: The Effect of Virtual Reality-Based Disaster Education Given to Nursing Students on Disaster Preparedness: Randomized Controlled Study
Brief Title: The Effect of Virtual Reality-Based Disaster Education Given to Nursing Students on Disaster Preparedness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: ZİYAFET UĞURLU (Unknown)
Responsible Party: Principal Investigator, Bekir Ertugrul, Lecturer, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BASKENTUNIVERSITY-001
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Disaster; Personality; Disorder, Mood
Keywords: Disaster; Disaster Preparedness; Psychological Preparedness; Nursing Students; Virtual Reality
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality (Experimental): The experimental group will be given virtual reality-based training in addition to standard training.
  Interventions: Behavioral: virtual reality
- standard training (No Intervention): The control group will be given only standard training.

INTERVENTIONS:
Behavioral: virtual reality — It is planned to provide 4 sessions of standard disaster preparedness training to nursing students in the intervention group. After the standard training sessions are completed, nursing students will be shown disaster simulation videos and visuals using virtual reality glasses within the scope of the virtual reality-based disaster preparedness training program.
  Arms: virtual reality

SUMMARY:
It is thought that, as a result of the virtual reality-based disaster training given to nursing students, the psychological preparedness of nursing students who will work before, during and after the disaster will increase in disaster preparedness and disaster threat. It is thought that this research will lead to the development of school-based interventions at other universities in similar situations.

The purpose of this research is to increase the level of psychological preparation and awareness of disaster preparedness and disaster threat through virtual reality-based disaster education given to nursing students.

ELIGIBILITY:
Inclusion Criteria:

* Being a 3rd and 4th year nursing student at the relevant universities where the study will be conducted,
* Not having taken the disaster management course before,
* Not having any health problems related to vision and hearing,
* Not wearing glasses to be able to use virtual reality (VR) glasses

Exclusion Criteria:

* Having any problems with vision or hearing
* Using glasses

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 67 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2024-04-29 (Actual)

PRIMARY OUTCOMES:
DİSASTER PREPARATION | 1-2 mounth
  Disaster preparedness level will be evaluated with the Disaster Threat Preparedness and Psychological Preparedness Scale. The minimum score that can be obtained from the scale is 13 and the maximum score is 52. As the score obtained from the scale increases, readiness also increases.

CONTACTS AND LOCATIONS:
Overall Officials: Bekir ERTUĞRUL, Principal Investigator — bertugrul@baskent.edu.tr
Locations (1):
- Başkent University, Ankara, Turkey (Türkiye)